CLINICAL TRIAL: NCT06516393
Title: Can Kinesio Tape Negatively Affect the Treatment by Creating a Hard Floor in Plantar Fasciitis Treatment: A Randomized Clinical Trial
Brief Title: Kinesio Tape Application in the Treatment of Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bihter Aslanyurek (Other)
Responsible Party: Sponsor-Investigator, Bihter Aslanyurek, associate professor, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEAH
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fasciitis; Radial Extracorporeal Shock Wave Therapy; Kinesio Taping; Pain
MeSH Terms: conditions — Fasciitis, Plantar; Pain

STUDY DESIGN:
Intervention Model Description: the patients were divided into subgroups by the sports physician according to age, height, body weight and body mass index. Patients with similar characteristics were randomized to one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radial extracorporeal shock wave therapy (r-ESWT) application group (Experimental): Patients with unilateral PF, that were randomly assigned into two groups receiving four sessions of either r-ESWT or r-ESWT+KT treatment once per week. All patients performed home exercises.
  Interventions: Device: The radial shock wave device
- r-ESWT + Kinesio taping (KT) application group (Active Comparator): Patients with unilateral PF, that were randomly assigned into two groups receiving four sessions of either r-ESWT or r-ESWT+KT treatment once per week. All patients performed home exercises.
  Interventions: Device: The radial shock wave device

INTERVENTIONS:
Device: The radial shock wave device — The r-ESWT+Kinesio Tape Application
  Other Names: The r-ESWT+Kinesio taping (KT)

SUMMARY:
This study is a prospective randomized clinical trial. Radial extracorporeal shock wave therapy (r-ESWT) is accepted as one of the most effective treatment modalities for plantar fasciitis (PF). Kinesio taping (KT) applied to the plantar fascia can provide patients with PF some benefits, but there no enough evidence about this topic. This study analysed the acute effect of adding KT to r-ESWT, on pain, foot function and flexibility when treating PF.

DETAILED DESCRIPTION:
The study was performed on 42 patients with unilateral PF, that were randomly assigned into wo groups receiving four sessions of either r-ESWT or r-ESWT+KT treatment once per week. All patients performed home exercises. Patients' pain levels were evaluated via the Visual Analogue Scale (VAS), and foot function via the Foot Function Index (FFI). Flexibility was assessed through gastro-soleus and plantar fascia flexibility tests. The evaluations were done before and one week after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral plantar fasciitis,
* The presence of a heel spur on a lateral radiograph

Exclusion Criteria:

* Lower extremity surgeries or traumas,
* Systemic inflammatory disease,
* Steroid injections administered within the past six months,
* Pacemaker usage,
* Coagulation disorders,
* Use of anticoagulants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the Visual Analog Scale (VAS) at week 5 | Baseline and week 5
  VAS is a tool where patients indicate the level of pain they feel using a 10 cm ruler. VAS pain score "no pain" (score=0) and "worst pain" (score=10).
Change from baseline Foot function via the Foot Function Index (FFI) at week 5 | Baseline and week 5
  FFI is a safe and valid foot-specific assessment measure used to evaluate pain, disability, and activity limitation, filled out by the patient self-reported
Change from baseline flexibility was evaluated through gastro-soleus and plantar fascia flexibility tests at week 5 | Baseline and week 5
  The patient was seated on a flat surface with the knees extended and the soles of the feet touching the wall. The tests were repeated three times and the average of the three measurements was taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Bihter Akınoğlu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once the study is published, data will be shared.
Access Criteria: If ethics committee requirements are met in similar studies to be conducted by clinical researchers, data can be shared with the permission of the clinical officer.

REFERENCES:
- [Derived] Kocahan T, Orscelik A, Gunaydin H, Buyukluoglu G, Karaaslan B, Asar E, Akinoglu B. Can kinesio tape negatively affect the treatment by creating a hard floor in plantar fasciitis treatment? A randomized clinical trial. PLoS One. 2025 May 5;20(5):e0322397. doi: 10.1371/journal.pone.0322397. eCollection 2025. PMID 40323967